CLINICAL TRIAL: NCT02320448
Title: Implementation and Evaluation of PIPAC for the Treatment of Patients With Peritoneal Carcinomatosis - a Feasibility Study.
Brief Title: Treating Peritoneal Carcinomatosis With PIPAC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Michael Bau Mortensen (Other)
Responsible Party: Sponsor-Investigator, Michael Bau Mortensen, Professor, Odense University Hospital
Organization: Odense University Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PIPAC
Record Dates: First submitted 2014-12-09; First posted 2014-12-19 (Estimated); Last update posted 2017-09-12 (Actual); Status verified 2017-09

CONDITIONS: Peritoneal Carcinomatosis
MeSH Terms: conditions — Peritoneal Neoplasms | interventions — Cisplatin; Doxorubicin; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- PIPAC (Experimental): PIPAC with cisplatin (7.5mg/m2 in 150 ml saline) and doxorubicin (1.5mg/m2 in 50 ml saline) in patients with peritoneal metastases (PM) from any origin besides colorectal/appendiceal cancers in whom oxaliplatin (92mg/m2 in 150 ml dextrose) will be used.
  The aerosolised chemotherapy will be nebulized at a flow of 0.5ml/min at a maximum pressure of 200 PSI during a standard laparoscopy with an intraabdominal pressure of 12mmHg. The CO2 will be evacuated 30 minutes after administration of chemotherapy and the patient is closed similar to a standard laparoscopy.
  Interventions: Drug: PIPAC

INTERVENTIONS:
Drug: PIPAC
  Other Names: Cisplatin; Doxorubicin; Oxaliplatin

SUMMARY:
This is a feasibility study that aims to evaluate whether PIPAC (Pressurized Intraperitoneal Aerosol Chemotherapy) is a safe and feasible treatment in Danish patients with peritoneal cancer.

DETAILED DESCRIPTION:
Peritoneal carcinomatosis (PC) represents end stage disease in many types of cancer (e.g. gastric, pancreatic, liver, colo-rectal, ovarian) and the majority of patients with PC will die from their disease within 6 months. Platinum-based systemic chemotherapy (SC) may prolong survival in selected patients, but poor performance status and low response rates have led to conservative (nihilistic) treatment strategies in these patients. However, patients with PC who are in good condition, and with a remaining life expectancy of more than a few months, may still have an unmet need for additional treatment in order to be able to perform with a high quality of life for as long as possible. These patients often have tried several lines of SC with disappointing results, and alternative and more effective treatment strategies are desperately needed.

The installation of chemotherapeutic agents within the peritoneal cavity would seem a simple and effective treatment of PC - at least from a theoretical point of view. Unfortunately, the effect of intraperitoneal chemotherapy on PC is disappointing. Like with SC, the poor response rates may be explained by the poor penetration of the active chemical substances into the PC plaques. Combining cytoreductive surgery (CRS) with intraperitoneal chemotherapy has gained interest in the recent years, but this approach can only be used in highly selected patients (where CRS is possible), and the procedure carries a significant risk of complications and side effects. Thus, a minimally invasive and safe delivery of relevant chemotherapy in such concentration that may allow it to work efficiently on the PC plaques would be an ideal platform for a new treatment strategy in these patients.

Pressurized IntraPeritoneal Aerosol Chemotherapy (PIPAC) Temperature and pressure are important factors during absorption of fluid from the peritoneal cavity, and the use of a relative low intraperitoneal pressure (2-6 mmHg) seems to increase the inflow of intraperitoneal fluid into the abdominal wall. Studies have confirmed that higher tissue concentrations of chemotherapy may be obtained by increasing the intraperitoneal pressure. After years of extensive testing, and the development of a micro-pump for safe aerosol infusion, a German research group has designed a system that allows a laparoscopy controlled, intraperitoneal aerosol infusion of chemotherapy (doxorubicin and cisplatin). The aerosol technique ensures that the entire peritoneal surface is covered by chemotherapy, and this is relevant in patients with PC. With the micro-pump positioned through a standard trocar pointing away from the bowels, a commercially available injection pump provides the necessary pressure to induce an aerosol mist covering the peritoneal cavity. After five minutes, the chemotherapy has been delivered, and the injector is turned off. After an additional 25 minutes of simple diffusion, the intra-abdominal air saturated with chemotherapy is evacuated through a standard trocar.

Recently, a German research group published their preliminary experience with PIPAC in gastric and ovarian cancer patients with PC .

PIPAC is not available freely on the market, and the procedure is not FDA approved yet. The German research team has emphasized, that despite the very encouraging results obtained so far, the efficacy and safety of PIPAC still has to be assessed in adequate clinical trials.

Aim In a compassionate use program, the aim of this study is to implement and evaluate the PIPAC procedure at Odense University Hospital under strict observation of both patient and occupational health safety aspects. Thus, it is important to emphasize, that the primary aim of this feasibility study is a quick and safe implementation of a new combined surgical-oncologic treatment technique which uses conventional chemotherapy in a new way in desperately ill cancer patients. For technical and safety reasons this implementation needs to be fulfilled and documented before patients can be enrolled in clinical trials.

Hypothesis The investigators expect the PIPAC procedure to be feasible and safe, with a primary non-access ratio of maximum 7:35 (mainly due to adhesions). The investigators expect a CTCAE grade of no more than 3 and that the procedure is safe for both patients, surgeons and OR staff.

Method

Study design This is a feasibility study where the PIPAC procedure will be performed in 35 patients fulfilling the inclusion criteria.

Implementation of the PIPAC procedure In order to cover all safety aspects and to secure optimal treatment results, a complete manual and checklist for the entire PIPAC procedure, as well as for pre- and postoperative patient handling, has been made. Thus, every step of the procedure is carefully described and monitored, and prior to the first patient treatment, the entire PIPAC procedure will be tried in a "dummy" OR setup supervised by the German group. Although this group has documented, that the procedure is safe for both patients and health care workers, the procedure will only be performed in an OR with laminar airflow and a closed carbon dioxide (CO2) ventilation system. In addition, environmental measurements (platinum particles within the OR) and bio-monitoring (blood samples) of the OR team are scheduled from the beginning of the first PIPAC procedure.

Preliminary clinical evaluation 35 patients with PC (see inclusion criteria) will be scheduled for PIPAC. In collaboration with the German group, the local multidisciplinary team (MDT) meeting will carefully select patients suitable for the PIPAC procedure. These patients are included according to national regulations and rules on experimental cancer research. All PIPAC procedures are performed with prophylactic antibiotics and start with a classification of the extent of the PC (Peritoneal Cancer Index, PCI) followed by selected quadrant biopsies to document malignancy and for later translational research. The type and doses of chemotherapy (1/10 of systemic dose), intra-abdominal pressure, temperature and delivery time are similar to those used by the German group. After the PIPAC procedure, the patients will be observed for two days before discharge. The treatment response is monitored by CT, and by a follow-up laparoscopy procedure with PCI score and biopsies after six weeks. The PIPAC procedure will be repeated during the same evaluation laparoscopy if objective response or no progression is observed. Adverse medical events will be graded according to the Common Terminology Criteria for Adverse Events (CTCAE, version 4.0), and surgical related complications according to the Dindo-Clavien classification.

Intra-abdominal access and completion of the PIPAC procedure in 28 of 35 patients and discharge of the same group within 2 POD are considered a successful implementation of the PIPAC procedure.

Occupational health safety aspects For safety reasons no staff is in the OR during the PIPAC procedure. The injector is controlled by a footswitch from outside the OR room, and observation monitors related to the anesthesiology are also made visible from outside the OR. Since no personnel are inside the ventilated OR room during application of the aerosolized chemotherapy, there are three barriers between surgeons/OR staff and the chemotherapy: The closed abdominal cavity, the laminar airflow system and the OR walls. The tightness of the abdominal cavity is controlled by allowing a maximum CO2 flow of 0.1-0.2 L/min corresponding to the body resorption of CO2. After the procedure, intraabdominal air saturated with chemotherapy is evacuated through a series of filters and into a closed system. Closure of the trocar sites, removal and disposal of dressings and syringes into special chemotherapy waste bins are performed by the surgeon alone. Environmental biomonitoring and blood samples from the surgeons and OR staff are scheduled as part of the safety monitoring.

Patient safety All patients are carefully selected (see exclusion criteria) on the MDT. The establishing of pneumoperitoneum and use of trocars are based on the highest standards for laparoscopic surgery which have a high safety profile. The procedures are performed by experienced laparoscopic surgeons under the supervision of the German team. When following the safety protocol used by the German group, no mortality related to the PIPAC procedure has been observed. The risk of bowel perforation is 2 per mille, port site metastases occur in 0.6% of the procedures, and self- limiting erythema around the trocar site is found in 1.2% of the procedures (private communication, professor Marc A. Reymond).

A short period of postoperative fever and/or elevated acute phase proteins have been observed after the PIPAC procedure, but the majority of patients may be discharged the same or the following day, and the PIPAC procedure can be repeated several times.

ELIGIBILITY:
Inclusion criteria

* Histological or cytological verified malignancy.
* Clinical or radiological evidence of peritoneal carcinomatosis.
* No indication for standard chemotherapy.
* Performance status 0-2 and life expectancy of more than 3 months.
* Age > 18 years.
* Written informed consent must be obtained according to the local Ethics Committee requirements.

Exclusion criteria

* Symptomatic small bowel obstruction (Total parenteral nutrition, nasogastric tube).
* Previous treatment with maximum cumulative doses of doxorubicin, daunorubicin, epirubicin, idarubicin, and/or other anthracyclines and anthracenediones.
* A history of allergic reaction to cisplatin or other platinum containing compounds or doxorubicin.
* Renal impairment, defined as GFR < 50 ml/min, (Cockcroft-Gault Equation).
* Myocardial insufficiency, defined as NYHA class > 2.
* Impaired liver function defined as bilirubin ≥ 1,5 x UNL (upper normal limit).
* Inadequate haematological function defined as ANC ≤ 1.5 x 109/l and platelets ≤ 100 x 109/l.
* Any other condition or therapy, which in the investigator's opinion may pose a risk to the patient or interfere with the study objectives.
* Previous intraabdominal chemotherapy or intraabdominal antibody therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Number of Patients with Adverse Events. | 5 months.
  No patients with adverse events above grade 3 on the CTCAE (Version 4) scale. No patients with complications above grade 2 on the Dindo-Clavien classification.

SECONDARY OUTCOMES:
Occupational health. | 5 months.
  No detectable chemotherapy on environmental biomonitoring and blood samples from the surgeons and OR staff.
Feasibility: Completion of procedure in 28:35 | 5 months.
  Completion of procedure in 28:35.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Mortensen, Professor, Study Director — Odense University Hospital
Locations (1):
- Odense University Hospital, Odense, Denmark

REFERENCES:
- [Background] Sugarbaker PH. Intraperitoneal chemotherapy and cytoreductive surgery for the prevention and treatment of peritoneal carcinomatosis and sarcomatosis. Semin Surg Oncol. 1998 Apr-May;14(3):254-61. doi: 10.1002/(sici)1098-2388(199804/05)14:33.0.co;2-u. PMID 9548609
- [Background] Coccolini F, Gheza F, Lotti M, Virzi S, Iusco D, Ghermandi C, Melotti R, Baiocchi G, Giulini SM, Ansaloni L, Catena F. Peritoneal carcinomatosis. World J Gastroenterol. 2013 Nov 7;19(41):6979-94. doi: 10.3748/wjg.v19.i41.6979. PMID 24222942
- [Background] Flessner MF. The transport barrier in intraperitoneal therapy. Am J Physiol Renal Physiol. 2005 Mar;288(3):F433-42. doi: 10.1152/ajprenal.00313.2004. PMID 15692055
- [Background] Dindo D, Demartines N, Clavien PA. Classification of surgical complications: a new proposal with evaluation in a cohort of 6336 patients and results of a survey. Ann Surg. 2004 Aug;240(2):205-13. doi: 10.1097/01.sla.0000133083.54934.ae. PMID 15273542
- [Result] Jacquet P, Stuart OA, Chang D, Sugarbaker PH. Effects of intra-abdominal pressure on pharmacokinetics and tissue distribution of doxorubicin after intraperitoneal administration. Anticancer Drugs. 1996 Jul;7(5):596-603. doi: 10.1097/00001813-199607000-00016. PMID 8862729
- [Result] Tempfer CB, Celik I, Solass W, Buerkle B, Pabst UG, Zieren J, Strumberg D, Reymond MA. Activity of Pressurized Intraperitoneal Aerosol Chemotherapy (PIPAC) with cisplatin and doxorubicin in women with recurrent, platinum-resistant ovarian cancer: preliminary clinical experience. Gynecol Oncol. 2014 Feb;132(2):307-11. doi: 10.1016/j.ygyno.2013.11.022. Epub 2013 Nov 23. PMID 24275155
- [Result] Solass W, Kerb R, Murdter T, Giger-Pabst U, Strumberg D, Tempfer C, Zieren J, Schwab M, Reymond MA. Intraperitoneal chemotherapy of peritoneal carcinomatosis using pressurized aerosol as an alternative to liquid solution: first evidence for efficacy. Ann Surg Oncol. 2014 Feb;21(2):553-9. doi: 10.1245/s10434-013-3213-1. Epub 2013 Sep 5. PMID 24006094
- [Result] Blanco A, Giger-Pabst U, Solass W, Zieren J, Reymond MA. Renal and hepatic toxicities after pressurized intraperitoneal aerosol chemotherapy (PIPAC). Ann Surg Oncol. 2013 Jul;20(7):2311-6. doi: 10.1245/s10434-012-2840-2. Epub 2013 Feb 3. PMID 23377563
- [Result] Solass W, Giger-Pabst U, Zieren J, Reymond MA. Pressurized intraperitoneal aerosol chemotherapy (PIPAC): occupational health and safety aspects. Ann Surg Oncol. 2013 Oct;20(11):3504-11. doi: 10.1245/s10434-013-3039-x. Epub 2013 Jun 14. PMID 23765417
- [Derived] Graversen M, Fristrup C, Kristensen TK, Larsen TR, Pfeiffer P, Mortensen MB, Detlefsen S. Detection of free intraperitoneal tumour cells in peritoneal lavage fluid from patients with peritoneal metastasis before and after treatment with pressurised intraperitoneal aerosol chemotherapy (PIPAC). J Clin Pathol. 2019 May;72(5):368-372. doi: 10.1136/jclinpath-2018-205683. Epub 2019 Feb 12. PMID 30755498
- [Derived] Graversen M, Detlefsen S, Bjerregaard JK, Fristrup CW, Pfeiffer P, Mortensen MB. Prospective, single-center implementation and response evaluation of pressurized intraperitoneal aerosol chemotherapy (PIPAC) for peritoneal metastasis. Ther Adv Med Oncol. 2018 Jun 1;10:1758835918777036. doi: 10.1177/1758835918777036. eCollection 2018. PMID 29899763